CLINICAL TRIAL: NCT01276951
Title: Controlled Clinical Trial of the Effect of Cocoa Consumption in Lowering Blood Pressure and in the Modulation of Endothelial Inflammation in Hypertensive Patients Assigned to an Entity Health Promoting.
Brief Title: Controlled Clinical Trial to Determine the Effective Dose of Cocoa in Lowering Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cacao III
Record Dates: First submitted 2010-05-24; First posted 2011-01-14 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Cocoa; Chocolate; Endothelial disfunction; Cardiovascular disease; Blood Pressure; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — Parturition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Delivery and return of chocolate; Procedure: Determination of blood pressure; Procedure: Anthropometric Measurements; Procedure: Food Anamnesis; Procedure: Samples: serological tests and culture of mononuclear cells; Procedure: Analysis of cytokine production
- 6,5g Dose Group (Active Comparator)
  Interventions: Dietary Supplement: Delivery and return of chocolate; Procedure: Determination of blood pressure; Procedure: Anthropometric Measurements; Procedure: Food Anamnesis; Procedure: Samples: serological tests and culture of mononuclear cells; Procedure: Analysis of cytokine production
- 12g Dose Group (Active Comparator)
  Interventions: Dietary Supplement: Delivery and return of chocolate; Procedure: Determination of blood pressure; Procedure: Anthropometric Measurements; Procedure: Food Anamnesis; Procedure: Samples: serological tests and culture of mononuclear cells; Procedure: Analysis of cytokine production
- 25g Dose Group (Active Comparator)
  Interventions: Dietary Supplement: Delivery and return of chocolate; Procedure: Determination of blood pressure; Procedure: Anthropometric Measurements; Procedure: Food Anamnesis; Procedure: Samples: serological tests and culture of mononuclear cells; Procedure: Analysis of cytokine production
- 50g Dose Group (Active Comparator)
  Interventions: Dietary Supplement: Delivery and return of chocolate; Procedure: Determination of blood pressure; Procedure: Anthropometric Measurements; Procedure: Food Anamnesis; Procedure: Samples: serological tests and culture of mononuclear cells; Procedure: Analysis of cytokine production

INTERVENTIONS:
Dietary Supplement: Delivery and return of chocolate — At baseline and then every 2 weeks, each participant will receive different grams of chocolate, according to the group to which he is assigned.
Procedure: Determination of blood pressure — Blood pressure will be determined at study entry, ninth and eighteenth week taking into account the protocols established in 2007 by the European Society of Cardiology and Hypertension. Because blood pressure has variations throughout the day and that measuring ambulatory health institutions can generate emotional changes that induce changes in this clinical setting, which for purposes of this study is the main outcome variable, there will be 24-hour monitoring of blood pressure at the beginning and end of the study.
Procedure: Anthropometric Measurements — The study will be determined the body mass index (BMI) by the ratio of weight in kilograms over height in meters squared, for which anthropometric measurement will be made at first, ninth and the eighteenth week as follows: The weight will be taken with an electronic balance of 0.05 g sensitivity standing capacity of 150 kg. We will be rated based on BMI cut points given by WHO-PAHO (1993) and adopted by the Ministry of Health of Colombia (2000).
Procedure: Food Anamnesis — With the aim of learning about the eating habits, it will be made based on a food intake recall the last 24 hours, taking into account that is not preceded by a special food day (sundays, holidays, celebrations). For more accurately calculate nutrient ingested food, modules will be used.
Procedure: Samples: serological tests and culture of mononuclear cells — At admission and at the end of the study will be obtained after 12 hours of fasting, 8 mL of blood in a dry tube without anticoagulant and 30 mL of blood in heparin tubes, properly labeled with the code assigned to the participant. The sample will be used to determine the complete lipid profile (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol and VLDL cholesterol), State of oxidation of low density lipoprotein (oxLDL) and mononuclear cell culture. The remaining serum was kept at -20°C for use if is required repeat any study.
Procedure: Analysis of cytokine production — We will be used the supernatant of mononuclears cell culture to quantify the production of interleukin one beta, interleukin two, tumor necrosis factor alpha by ELISA with commercially available kits for this purpose.

SUMMARY:
In Colombia, ischemic heart disease and stroke are one of the most important causes of death in 45 years old people. Care of cases of disease represents high costs for the health system in particular and society in general, due to the loss of productive years life and costs for the care of the aftermath. Hypertension (HT) is one of the preventable risk factors for major cerebrovascular disorders. The pathophysiology of Essential hypertension is complex and depends of interaction of genetic and environmental factors. Among the determining elements are the increase in the activity of the sympathetic nervous system, the vasoconstricting and overproduction of hormones associated with sodium retention, disruption in renin secretion with increased production of aldosterone and angiotensin II, the deregulation of the kinins system, the increase in peripheral vascular resistance and activity of Growth factors in atherogenesis and vascular endothelial dysfunction, increased cardiac output, diabetes mellitus, obesity, and lower production of vasodilators such as brain natriuretic peptide (BNP), the prostacyclins and nitric oxide (NO), among others.

Cocoa is a food rich in flavonoids, which stimulate the enzyme activity of endothelial nitric oxide synthase (e-NOS), responsible of the production of NO in vascular smooth muscle. The flavonoids modulate the synthesis of inflammatory substances that are derived from endothelial cells and the immune system.

In a recent study found that with a few grams of cocoa achieves a significant reduction in blood pressure, so the investigators propose a controlled clinical trial to assess the effect of different doses of cocoa on blood pressure and endothelial inflammation in men with essential hypertension, stage I-II without target organ damage, in addition to pharmacologic monotherapy defined for the management of their disease. The investigators hope to determine an optimal dose of cocoa, with long-term effects, by their high content of flavonoids, improves cardiovascular and endothelial parameters with the advantage that it is an economical and easy introduction into the patient's habits.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age: 18 - 65 years old
* Resides in Medellín City
* Attached from the contributive regimen of Colombian Health System
* Essential Arterial Hypertension, stage I or II.
* Be receiving pharmacologic therapy (maximum 2 medications), whose dose has been stable for eight weeks prior to study entry.
* Voluntary desire to consume 6,5; 12; 25 or 50 grams of chocolate per day for 18 weeks.
* Voluntary desire to participate in the trial and sign informed consent.

Exclusion Criteria:

* Secondary hypertension
* Injury in target organ: heart, kidney, brain and retina
* Presence of diabetes mellitus
* BMI (Body Mass Index) major or equal to 30
* Present smoker or with less than four weeks of abstinence of tobacco
* Consume antiplatelet substances
* Regular consumption of antioxidants and multivitamins
* During the study excluded any participant to present a sudden increase in blood pressure: SBP greater than or equal to 180 mmHg and/or DBP greater or equal to 110 mm Hg.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change on blood pressure in patients with stage I-II hypertension, after consumption of different doses of cocoa. | 18 weeks

SECONDARY OUTCOMES:
Change in the oxidation of low density lipoproteins after cocoa consumption, in patients with stage I-II hypertension. | 18 weeks
Change in the production of inflammatory molecules derived from peripheral blood mononuclear cells of patients with arterial hypertension stage I-II, after cocoa consumption. | 18 weeks
Change in platelet aggregation after cocoa consumption, in patients with essential arterial hypertension stage I-II. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mónica L. Giraldo Restrepo, Nurse. PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Sede Investigaciones Universitarias, Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grassi D, Necozione S, Lippi C, Croce G, Valeri L, Pasqualetti P, Desideri G, Blumberg JB, Ferri C. Cocoa reduces blood pressure and insulin resistance and improves endothelium-dependent vasodilation in hypertensives. Hypertension. 2005 Aug;46(2):398-405. doi: 10.1161/01.HYP.0000174990.46027.70. Epub 2005 Jul 18. PMID 16027246
- [Background] WHO publishes definitive atlas on global heart disease and stroke epidemic. Indian J Med Sci. 2004 Sep;58(9):405-6. No abstract available. PMID 15902773
- [Background] Oparil S, Zaman MA, Calhoun DA. Pathogenesis of hypertension. Ann Intern Med. 2003 Nov 4;139(9):761-76. doi: 10.7326/0003-4819-139-9-200311040-00011. No abstract available. PMID 14597461
- [Background] Cifkova R. The burden of hypertension and inadequate control in populations. J Hypertens. 2006 May;24(5):807-9. doi: 10.1097/01.hjh.0000222745.52325.e7. No abstract available. PMID 16612237
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Kearney PM, Whelton M, Reynolds K, Whelton PK, He J. Worldwide prevalence of hypertension: a systematic review. J Hypertens. 2004 Jan;22(1):11-9. doi: 10.1097/00004872-200401000-00003. PMID 15106785
- [Background] Aristizabal D GE, McEwen J, Caulfiel M, Mendez J, Medina E, Zapata N, Correa M. Bases genéticas de la hipertension arterial esencial en Colombia: avances en nueve años de estudio. Revista Colombiana de Cardiología. 12(6), 2006.
- [Background] Beevers G, Lip GY, O'Brien E. ABC of hypertension: The pathophysiology of hypertension. BMJ. 2001 Apr 14;322(7291):912-6. doi: 10.1136/bmj.322.7291.912. No abstract available. PMID 11302910
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A, Vahanian A, Camm J, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Erdine S, Kiowski W, Agabiti-Rosei E, Ambrosioni E, Lindholm LH, Viigimaa M, Adamopoulos S, Agabiti-Rosei E, Ambrosioni E, Bertomeu V, Clement D, Erdine S, Farsang C, Gaita D, Lip G, Mallion JM, Manolis AJ, Nilsson PM, O'Brien E, Ponikowski P, Redon J, Ruschitzka F, Tamargo J, van Zwieten P, Waeber B, Williams B; Management of Arterial Hypertension of the European Society of Hypertension; European Society of Cardiology. 2007 Guidelines for the Management of Arterial Hypertension: The Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2007 Jun;25(6):1105-87. doi: 10.1097/HJH.0b013e3281fc975a. No abstract available. PMID 17563527
- [Background] Steinberg D. Atherogenesis in perspective: hypercholesterolemia and inflammation as partners in crime. Nat Med. 2002 Nov;8(11):1211-7. doi: 10.1038/nm1102-1211. No abstract available. PMID 12411947
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Taubert D, Roesen R, Schomig E. Effect of cocoa and tea intake on blood pressure: a meta-analysis. Arch Intern Med. 2007 Apr 9;167(7):626-34. doi: 10.1001/archinte.167.7.626. PMID 17420419
- [Background] Schroeter H, Heiss C, Balzer J, Kleinbongard P, Keen CL, Hollenberg NK, Sies H, Kwik-Uribe C, Schmitz HH, Kelm M. (-)-Epicatechin mediates beneficial effects of flavanol-rich cocoa on vascular function in humans. Proc Natl Acad Sci U S A. 2006 Jan 24;103(4):1024-9. doi: 10.1073/pnas.0510168103. Epub 2006 Jan 17. PMID 16418281
- [Background] McCullough ML, Chevaux K, Jackson L, Preston M, Martinez G, Schmitz HH, Coletti C, Campos H, Hollenberg NK. Hypertension, the Kuna, and the epidemiology of flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S103-9; discussion 119-21. doi: 10.1097/00005344-200606001-00003. PMID 16794446
- [Background] Fisher ND, Sorond FA, Hollenberg NK. Cocoa flavanols and brain perfusion. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S210-4. doi: 10.1097/00005344-200606001-00017. PMID 16794460
- [Background] Tsuruchi N, Jimi S. [A case of recurrent endometrial cancer successfully treated with oral administration of etoposide]. Gan To Kagaku Ryoho. 1992 Jan;19(1):103-5. Japanese. PMID 1729957
- [Background] Farouque HM, Leung M, Hope SA, Baldi M, Schechter C, Cameron JD, Meredith IT. Acute and chronic effects of flavanol-rich cocoa on vascular function in subjects with coronary artery disease: a randomized double-blind placebo-controlled study. Clin Sci (Lond). 2006 Jul;111(1):71-80. doi: 10.1042/CS20060048. PMID 16551272
- [Background] Taubert D, Roesen R, Lehmann C, Jung N, Schomig E. Effects of low habitual cocoa intake on blood pressure and bioactive nitric oxide: a randomized controlled trial. JAMA. 2007 Jul 4;298(1):49-60. doi: 10.1001/jama.298.1.49. PMID 17609490
- [Background] Taubert D, Berkels R, Roesen R, Klaus W. Chocolate and blood pressure in elderly individuals with isolated systolic hypertension. JAMA. 2003 Aug 27;290(8):1029-30. doi: 10.1001/jama.290.8.1029. No abstract available. PMID 12941673
- [Background] Grassi D, Lippi C, Necozione S, Desideri G, Ferri C. Short-term administration of dark chocolate is followed by a significant increase in insulin sensitivity and a decrease in blood pressure in healthy persons. Am J Clin Nutr. 2005 Mar;81(3):611-4. doi: 10.1093/ajcn/81.3.611. PMID 15755830
- [Background] Heiss C, Dejam A, Kleinbongard P, Schewe T, Sies H, Kelm M. Vascular effects of cocoa rich in flavan-3-ols. JAMA. 2003 Aug 27;290(8):1030-1. doi: 10.1001/jama.290.8.1030. No abstract available. PMID 12941674
- [Background] Mursu J, Voutilainen S, Nurmi T, Rissanen TH, Virtanen JK, Kaikkonen J, Nyyssonen K, Salonen JT. Dark chocolate consumption increases HDL cholesterol concentration and chocolate fatty acids may inhibit lipid peroxidation in healthy humans. Free Radic Biol Med. 2004 Nov 1;37(9):1351-9. doi: 10.1016/j.freeradbiomed.2004.06.002. PMID 15454274
- [Background] Binder CJ, Chang MK, Shaw PX, Miller YI, Hartvigsen K, Dewan A, Witztum JL. Innate and acquired immunity in atherogenesis. Nat Med. 2002 Nov;8(11):1218-26. doi: 10.1038/nm1102-1218. No abstract available. PMID 12411948
- [Background] Selmi C, Mao TK, Keen CL, Schmitz HH, Eric Gershwin M. The anti-inflammatory properties of cocoa flavanols. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S163-71; discussion S172-6. doi: 10.1097/00005344-200606001-00010. PMID 16794453
- [Background] Keen CL, Holt RR, Oteiza PI, Fraga CG, Schmitz HH. Cocoa antioxidants and cardiovascular health. Am J Clin Nutr. 2005 Jan;81(1 Suppl):298S-303S. doi: 10.1093/ajcn/81.1.298S. PMID 15640494